CLINICAL TRIAL: NCT01503983
Title: Phase II Study to Assess the Efficacy and Safety of Trastuzumab in Combination With Xelox as First-line Treatment of Patients With Advanced or Metastatic Gastric Cancer or Gastro-esophageal Junction, (HER2)-Positive.
Brief Title: Efficacy and Safety of Trastuzumab, Capecitabine y Oxaliplatine as Treatment Gastric Cancer Metastatic (HER2)Positive
Acronym: HerXO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación para el Progreso de la Oncología en Cantabria (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUPOCAN-01-11; 2011-001231-23 (EudraCT Number)
Record Dates: First submitted 2011-12-07; First posted 2012-01-04 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2012-04

CONDITIONS: Stage IV Gastric Cancer With Metastasis
Keywords: Gastric Cancer with Metastasis; HER2-positive
MeSH Terms: interventions — Trastuzumab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trastuzumab+Oxaliplatine+capecitabine (Experimental): Patient takes Trastuzumab (initial dose 8 mg/kg and a maintenance dose 6 mg/kg) anda oxaliplatin (dose 130mg/m2) during the first day os cycle and them Capecitabine (dose 2000 mg/m2)during 14 days in cycle of 21 days.
  Interventions: Drug: Trastuzumab; Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab: 8 mg/kg day 1 followed by 6 mg/kg every 3 weeks (i.v.)
  Other Names: Herceptin
Drug: Capecitabine — Capecitabine: 1000 mg/m2/12h/days 1 - 14 every 3 weeks (v.o.)
  Other Names: Xeloda
Drug: Oxaliplatin — Oxaliplatin: 130 mg/m2 in 2 h, day 1 / (i.v.) /every 3 weeks
  Other Names: Oxaliplatino

SUMMARY:
The objective of the study is assess the efficacy and safety of Trastuzumab in combination with Capecitabine+Oxaliplatin as first-line treatment of patients with advanced or metastatic gastric cancer or gastro-esophageal junction, (HER2)-positive.

DETAILED DESCRIPTION:
Gastric cancer worldwide is the second tumor incidence (10%). There are significant geographical differences in Spain with an incidence of 15 cases/100,000 per year. Although the incidence and mortality of gastric cancer (GC) have experienced a marked reduction in the past 40 years, this disease remains a leading cause of cancer-related mortality, accounting for more than 870,000 deaths worldwide in the year 2000.

Gastric cancer has a high mortality rate because usually diagnosed when in advanced stage and in many cases has a high relapse rate. Advanced gastric cancer cases are considered to be diagnosed with unresectable disease, either by having locally advanced disease (30% of cases at diagnosis), or having metastatic disease (another 30%) and patients with relapses (60% of resected). Thus, overall around 84% of patients with gastric cancer will have advanced disease.

The only curative treatment so far is surgery. Thanks to early detection and implementation of appropriate surgical techniques, survival has improved in some countries such as Japan and Korea, being the rate of 5-year survival of 47%Over the years, a large number of studies with a single agent chemotherapy has been shown that gastric cancer is a relatively sensitive to chemotherapy. Based on these observations, the trend was the investigation of the combination of chemotherapy agents.

Based on these results FDA and EMEA has approved capecitabine in the treatment of advance gastric cancer combined with platinum.

ELIGIBILITY:
Inclusion Criteria:

* Patients be able to grant a written informed consent or oral consent
* Age ≥18 years old
* Patients diagnosed with metastatic gastric or gastro-esophageal junction adenocarcinoma (HER2-positive), unresectable and histologically confirmed Measurable disease, following the new RECIST criteria,
* HER2 positive tumors (primary or metastatic) with overexpression HER2 determinated by IHQ +++ (IHQ3+) o IHQ ++ confirmed by FISH/SISH positive (IHQ2+/FISH+)
* ECOG ≤ 2
* Patients of childbearing potential (< 12 months from last menstruation), they have to use effective means of contraception
* Life expectancy more than 3 months
* Adequate renal function: calculated creatinine clearance > 50 mL/min
* Adequate liver function: AST and ALT ≤2.5 x LSN (5 x LSN with liver metastasis), bilirubin 1,5 x LSN. alkaline phosphatase < 2,5 x LSN (≤ 5 x LSN with liver metastasis o < 10 x LSN with bone metastases Adequate haematological function: Hb ≥9 g/dl, neutrophils ≥ 1,5 x 109 /l and platelets 100 x 109 /l.
* Normal Left Ventricle Fraction Ejection , LVEF> 50%
* Every patient should be treated and followed in his / her study site

Exclusion Criteria:

* Prior chemotherapy treatment for advanced/metastatic disease
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption
* Patients with active gastrointestinal bleeding
* Prior chemotherapeutic treatment for advanced / metastatic disease
* Toxicity as a result of prior therapy (except alopecia)., for example.
* Neurology toxicity grade ≥2NCI-CTCAE
* Patients who received radiotherapy within 4 weeks prior to study treatment.
* Major surgical procedures within 4 weeks prior to treatment without a total surgical recovery.
* Past or current history of other malignancies (within the last 5-2 years prior to treatment start), patients with curatively treated basal cell carcinoma of the skin or in situ carcinoma of the cervix are eligible
* Active and clinically significant cardiovascular disease,
* History or current clinical evidence of brain metastasis
* Patients undergoing transplantation allogenic requiring immunosuppressive treatment
* Moderate or severe renal failure, creatinine clearance < 50 mL/min, calculated by Cockcroft-Gault
* Adequate liver function: bilirubin ≤1.5 x UL, GOT ( ASAT )/ GPT ( ALAT ) ≤2,5 LSN. Liver metastasis ≤ 5 x LSN, FA ≤ de 2,5 feces el LSN.
* Adequate haematology function: neutrophils ≥ 1,5 x 109 /l and platelets 100 x 109 /l
* Treatment with sorivudine and the analogous as brivudine.
* Dihydropyrimidine proven dehydrogenase deficiency (DPD).
* Patients who had received any drug, agent or investigational procedure, or who have participated in another research study within 30 days prior to initiation of treatment with study medication.
* Hypersensitivity to any of the study drugs
* Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment-related complications
* Patients receiving chronic corticosteroid therapy or high dose (is allowed to use inhaled steroids and cycle short treatment with oral steroids for prevention of emesis or to stimulate appetite)
* Pregnancy and lactation
* Patients of childbearing potential not willing to use effective means of contraception.
* History of psychiatric disorders that the investigator considered clinically significant, causing the patient give informed consent or interfere with compliance with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-08; Primary Completion 2013-12 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Overall Survival | up to 10 Months
  Overall survival defined as the time from start of treatment until the patient's death

SECONDARY OUTCOMES:
progression free survival | 5 months
  Progression free survival defined as time from start of treatment until date of progression were observed according to RECIST 1.1
the time to progression | 5 months
  Time to progression defined as time elapsed since the beginning of treatment until disease progression
duration of response | 10 months
  Duration of response defined as the time since the objective complete or partial response until there is disease progression
time to response | 10 months
  Time to response, defined as the time from initiation of treatment until objective complete or partial response

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Rivera NA, Doctor, Principal Investigator — Sponsor represntative
Locations (13):
- Spain (13):
  - Hospital Juan Canalejo, A Coruña, A Coruña
  - Centro Oncológico de Galicia, A Coruña, A Coruña
  - Hospital Lucus Augusti de Lugo, Lugo, A Coruña
  - Hospital de Basurto, Bilbao, Bilbao
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Arnau de Vilanova de LLeida, Lleida, Lleida
  - Hospital Gregorio Marañon, Madrid, Madrid
  - Hospital La Paz, Madrid, Madrid
  - Hospital de Orense, Ourense, Orense
  - Hospital Universitario Cnetral de Asturias, Oviedo, Oviedo
  - Hospital Provincial de Pontevedra, Pontevedra, Vigo
  - Hospital Xeral Cies, Vigo, Vigo
  - Hospital de POVISA, Vigo, Vigo